CLINICAL TRIAL: NCT05455996
Title: An Open Label Study to Treat Post-Traumatic Stress in COVID-19 Healthcare Workers Using MDMA-Assisted Therapy
Brief Title: MDMA-Assisted Therapy for Stress Disorders in Healthcare Workers
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nautilus Sanctuary (Other)
Collaborators: Nautilus Psychiatric Services, PLLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSCF1/NSCovid-1
Record Dates: First submitted 2022-07-10; First posted 2022-07-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Post-Traumatic Stress Disorder; Adjustment Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Adjustment Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Single-arm, open label study to treat symptoms of Post-Traumatic Stress in 30 Health Care Workers using a 3-dosing model of MDMA-assisted therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MDMA-assisted therapy (Experimental): Participants will receive 3-dosing model of MDMA-assisted therapy (includes 9 non-drug therapy sessions)
  Interventions: Drug: MDMA

INTERVENTIONS:
Drug: MDMA — MDMA-assisted therapy
  Other Names: MDMA-assisted therapy

SUMMARY:
The purpose of this study is to assess the safety and efficacy of MDMA-Assisted Therapy on Health Care Workers suffering from symptoms of Post-Traumatic Stress due to their work on the frontline of the COVID Pandemic.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, screening participants who sign the Informed Consent form will go through multiple screening visits (onsite and remote) designed to assess psychiatric and medical appropriateness for the study treatment. Tapering of certain medications are required. The screening period takes between 3 to 7 weeks and includes two preparatory sessions (90 minutes each) with the participant's assigned therapy team.

Once a screening participant is deemed eligible for the study, baseline measures of symptomatology are obtained and a third preparatory session is conducted. The participant then enters into the Active Treatment Period which begins with the first of three all-day dosing sessions followed by three 90-minute integration (non-drug) sessions scheduled approximately a week and a half apart. Approximately 3 to 5 weeks after the first dosing session, a second all-day dosing session takes place, followed again by three 90-minute integration (non-drug) sessions scheduled about a week and a half apart. Approximately 3 to 5 weeks after the second dosing session, a third all-day dosing session takes place, followed again by three 90-minute integration (non-drug) sessions scheduled about a week and a half apart. The total time to complete the Active Treatment Phase is between 6 and 16 weeks.

Two to four weeks after the Active Treatment Phase, participants will meet with therapy team for a Treatment Termination Visit during which participants will complete primary outcome measures. Twelve months later, participants will be contacted and asked to repeat study measures to assess durability of effects.

From Screening to Treatment Termination, participation in the study takes between 11 and 33 weeks. Some non-drug sessions can be done remotely at the discretion of the therapy team.

ELIGIBILITY:
Inclusion Criteria:

* Were exposed to stressors related to their work in a health care setting during the COVID-19 pandemic
* Live full-time within a 60-mile radius of New York City.
* Are fluent in speaking and reading English.
* Are able to swallow pills.
* Agree to have study visits recorded, including Experimental Sessions, and non-drug therapy sessions.
* Have a contact (relative, spouse, close friend or other Support Person) who is willing and able to be reached by the Sponsor-Investigators in the event of a participant becoming suicidal or unreachable.
* Agree to inform the Sponsor-Investigators within 48 hours of any medical conditions and procedures.
* If able to become pregnant, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session.
* Comply with requirements for fasting and refraining from certain medications prior to Experimental Sessions, not participate in any other interventional clinical trials during the duration of the study, be driven home after Experimental Sessions, and commit to medication dosing, therapy, and study procedures.

Exclusion Criteria:

* Have previously participated in a clinical treatment trial using MDMA.
* Have a past diagnosis of PTSD unrelated to the COVID-19 pandemic.
* Have received Electroconvulsive Therapy (ECT) within 12 weeks of enrollment.
* Have a history of or a current primary psychotic disorder or bipolar I disorder
* Have a current eating disorder with active purging
* Have current major depressive disorder with psychotic features
* Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate
* Have uncontrolled essential hypertension
* Have a history of ventricular arrhythmia at any time, other than premature ventricular contractions (PVCs) in the absence of ischemic heart disease.
* Have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation.
* Have a history of arrhythmia, other than premature atrial contractions (PACs) or occasional PVCs in the absence of ischemic heart disease, within 12 months of screening.
* Have a marked Baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] in males and >460 ms in females corrected by Fridericia's formula).
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Require use of concomitant medications that prolong the QT/QTc interval during Experimental Sessions.
* Have symptomatic liver disease or have significant liver enzyme elevations.
* Have a history of hyponatremia or hyperthermia.
* Weigh less than 48 kilograms (kg).
* Are pregnant or nursing, or able to become pregnant and are not practicing an effective means of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on symptoms of Post-Traumatic Stress based on the PTSD Checklist for DSM-5 (PCL-5) at Treatment Termination | Up to 17 weeks post-enrollment (Baseline)
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD and is widely used by researchers and clinicians to monitor change during and after a treatment intervention. Participants indicate how much distress they have experienced due to symptoms such as "Repeated, disturbing memories, thoughts, or images of a stressful experience from the past," "Trouble remembering important parts of a stressful experience from the past," and "Feeling irritable or having angry outbursts" using a Likert scale ranging from 0 (Not at all) to 4 (Extremely). Items are summed to provide a total severity score (range = 0-80). It takes 5-10 minutes to complete.

SECONDARY OUTCOMES:
Change from Baseline on symptoms of Adjustment Disorder based on the Adjustment Disorder New Module-20 (ADNM-20) at Treatment Termination | Up to 17 weeks post-enrollment (Baseline)
  The ADNM-20 is a 20-item self-report questionnaire that measures AjD symptomatology and has two parts. In the first part, participants go through a list of typical stressors, mark the presence and timing of any that apply, and indicate the one stressor that was the most straining. In the second part, the participant ranks using a 4-point Likert scale, ranging from 1 (never) to 4 (often) the degree to which the most significant stressor may be causing troublesome reactions. The ADNM-20 consists of six subscales: preoccupation (4 items), failure to adapt (4 items), avoidance (4 items), depressive mood (3 items), anxiety (2 items), and impulse disturbance (3 items). ). It takes 5-10 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Willa Hall, Ph.D., Study Director — Nautilus Sanctuary; Casey Paleos, M.D., Principal Investigator — InnerMost PBC
Locations (2):
- United States (2):
  - Memoru, Boulder, Colorado
  - InnerMost, PBC, New York, New York

IPD SHARING:
Plan to Share IPD: No